CLINICAL TRIAL: NCT00033384
Title: A Multicenter Phase 2 Study of CI-1040 In Patients With Advanced Nonsmall-Cell Lung Cancer, Breast Cancer, Colon Cancer Or Pancreatic Cancer
Brief Title: CI-1040 in Treating Patients With Advanced Breast, Colon, Pancreatic, or Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000069279; UAB-0152; PFIZER-1040-002-004; UAB-F011203011; NCI-G02-2052
Record Dates: First submitted 2002-04-09; First posted 2003-07-08 (Estimated); Last update posted 2013-04-12 (Estimated); Status verified 2002-12

CONDITIONS: Breast Cancer; Colorectal Cancer; Lung Cancer; Pancreatic Cancer
Keywords: stage III colon cancer; stage IV colon cancer; stage IV breast cancer; stage IIIA breast cancer; recurrent breast cancer; stage IIIB breast cancer; recurrent non-small cell lung cancer; stage II pancreatic cancer; stage III pancreatic cancer; recurrent pancreatic cancer; recurrent colon cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; duct cell adenocarcinoma of the pancreas; stage IV pancreatic cancer
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Lung Neoplasms; Pancreatic Neoplasms; Colonic Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — 2-(2-chloro-4-iodophenylamino)-N-cyclopropylmethoxy-3,4-difluorobenzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: CI-1040

SUMMARY:
RATIONALE: CI-1040 may stop the growth of tumors by blocking the enzymes necessary for cancer cell growth and by stopping blood flow to the tumor.

PURPOSE: Phase II trial to study the effectiveness of CI-1040 in treating patients who have metastatic or unresectable breast, colon, pancreatic, or non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the antitumor activity of CI-1040 in patients with non-small cell lung, breast, colon, or pancreatic cancer.
* Determine the safety profile of this drug in these patients.
* Assess quality of life (overall and for each tumor type) of patients treated with this drug.
* Determine the relationship between study drug concentration and antitumor response in these patients and target suppression and safety of this drug.
* Correlate target suppression (pERK) with antitumor effects of this drug in these patients.
* Correlate the mRNA expression profile of the tumors with antitumor effects of this drug in these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to tumor type (non-small cell lung vs breast vs colon vs pancreas).

Patients receive oral CI-1040 twice daily on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline and then every 28 days during the first 6 months of study therapy.

Patients are followed every 2 months.

PROJECTED ACCRUAL: A total of 52-172 patients (13-43 per stratum) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed metastatic or inoperable non-small cell lung, breast, or colon cancer or duct cell carcinoma of the exocrine pancreas
* Bidimensionally measurable lesions that are not previously irradiated

  * New lesions that have developed in a previously irradiated field may be used as measurable disease
* No brain metastases

  * Patients with prior brain metastases are allowed provided they have undergone prior resection of metastases and/or 1 prior course of cranial irradiation, have no new sites of brain metastases since then, have no worsening CNS symptoms, and have discontinued prior corticosteroids for at least 30 days
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Not specified

Menopausal status:

* Not specified

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 2 times upper limit of normal (ULN)
* AST or ALT no greater than 2 times ULN (5 times ULN if due to liver involvement)

Renal:

* Creatinine no greater than 1.5 times ULN

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 30 days after study participation
* Capable of swallowing intact study medication capsules
* Capable of following instructions regarding study medication or has daily caregiver to administer study medication
* No concurrent serious infection
* No life-threatening illness unrelated to tumor
* No other prior or concurrent malignancy within the past 3 years except nonmelanoma skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 2 weeks since prior immunotherapy or biologic therapy

Chemotherapy:

* At least 4 weeks since prior cytotoxic chemotherapy
* No more than 1 prior cytotoxic chemotherapy regimen for metastatic non-small cell lung or colon cancer
* No more than 2 prior cytotoxic chemotherapy regimens for breast cancer
* No prior cytotoxic chemotherapy for pancreatic cancer

Endocrine therapy:

* See Disease Characteristics
* At least 2 weeks since other prior hormonal therapy

Radiotherapy:

* See Disease Characteristics
* At least 3 weeks since prior radiotherapy and recovered
* No concurrent radiotherapy

Surgery:

* See Disease Characteristics

Other:

* No other concurrent anticancer agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-02; Primary Completion 2003-11 (Actual); Study Completion 2003-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John J. Rinehart, MD, Study Chair — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama, United States